CLINICAL TRIAL: NCT04238247
Title: Tiny Cargo, Big Deal! An Adaptive ED-Based eHealth Intervention to Promote Correct and Consistent Size-Appropriate Child Passenger Safety Behaviors and Reduce Disparities
Brief Title: Tiny Cargo, Big Deal! An ED-Based Study of Child Passenger Safety Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Michelle Macy, MD, Director, Mary Ann & J. Milburn Smith Child Health Outcomes, Research, and Evaluation Center, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HD092594
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Accident, Traffic
Keywords: child restraint systems (car seats and booster seats); seat belts; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: After the baseline survey, all participants will be randomized into one of two groups: 1) basic intervention or 2) control group. Block randomization (block sizes from four to eight) will be applied to assign participants to intervention or control in a 3:1 ratio. Blocks will be stratified by child passenger safety recommendations for age (<2 years, rear-facing; 2-4 years, forward-facing; 5+ years, booster seat) and reason for study eligibility (not consistently using the recommended restraint for age and size or planning a premature transition in the coming 6 months).
  After 6-month follow-up, participants in the intervention group only who continue suboptimal child passenger safety behaviors will be re-randomized in a 1:1 ratio to basic or enhanced intervention.
Who Masked: Outcomes Assessor
Masking Description: This is a single-blinded study where a portion of the study will include blinding of study team members who are assessing outcomes. The blinding will not include the participants.
  The portion of the study that includes blinding is the review of the monthly photo submissions. Participants send us via text message over the course of 12 months. Each photograph is reviewed and scored by two team members. The first reviewer is blinded to study condition and saves the photographs with the child's face blurred. The second reviewer scores the photographs after the child's face has been blurred to verify findings of the first reviewer. The second reviewer is then unblinded to send feedback to the caregiver appropriate for their study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Usual Care (No Intervention): Participants will be randomized after completion of the baseline survey and receive a basic information sheet (print or electronic).
  Months 1-12: Participants receive monthly, unscheduled requests to submit photographs as their child usually travels. Feedback is provided for critical errors and misuse. Follow-up occurs at 6 months. Outcomes are assessed at 12 months.
- Basic Intervention (Experimental): Participants will be randomized after completion of the baseline survey and receive a basic information sheet (print or electronic). Participants receive a counseling session, access to the study's tailored, educational website, and tailored informational and motivational text messages.
  Months 1-6: Participants receive monthly, unscheduled requests to submit photographs as their child usually travels. Feedback is provided. Follow-up occurs at 6 months.
  After completion of their 6 month follow-up, participants in the Basic Intervention group will be eligible for re-randomization if they continue to not adhere to guidelines or plan a premature transition.
  Months 7-12: Participants continue to receive monthly, unscheduled requests to submit photographs as their child usually travels. Feedback is provided. Outcomes are assessed at 12 months.
  Interventions: Behavioral: Tiny Cargo, Big Deal/Abróchame Bien, Cuídame Bien (TCBD/ABCB) Basic Intervention
- Enhanced Intervention (Experimental): After completion of their 6 month follow-up, participants re-randomized to Enhanced Intervention receive Basic Intervention components plus an additional counseling session (Months 7/8) and additional tailored text messages (Months 7-12).
  Months 7-12: Participants continue to receive monthly, unscheduled requests to submit photographs as their child usually travels. Feedback is provided. Outcomes are assessed at 12 months.
  Interventions: Behavioral: Tiny Cargo, Big Deal/Abróchame Bien, Cuídame Bien (TCBD/ABCB) Basic Intervention; Behavioral: Tiny Cargo, Big Deal/Abróchame Bien, Cuídame Bien (TCBD/ABCB) Enhanced Intervention

INTERVENTIONS:
Behavioral: Tiny Cargo, Big Deal/Abróchame Bien, Cuídame Bien (TCBD/ABCB) Basic Intervention — A bilingual emergency department (ED)-based precision prevention intervention grounded in Self-Determination Theory. The Basic TCBD/ABCB intervention integrates one personalized counseling session based on principles of motivational interviewing (MI) and eHealth components including a tailored mobile-friendly educational website and short message service (SMS) text message communications with the goal of improving child passenger safety.
  Participants receive monthly text message requests to submit photographs depicting the child as they usually travel. Feedback is provided via text message to correct any observed errors or misuse. Tailored informational and motivational text messages are sent twice each month.
  Arms: Basic Intervention; Enhanced Intervention
Behavioral: Tiny Cargo, Big Deal/Abróchame Bien, Cuídame Bien (TCBD/ABCB) Enhanced Intervention — The Enhanced TCBD/ABCB Intervention includes a second motivational interviewing session. Basic Intervention text messages continue with an additional 1-2 tailored text messages per month.
  Arms: Enhanced Intervention

SUMMARY:
This study involves an emergency department (ED)-based intervention utilizing Motivational Interviewing (MI) techniques and patient-centered eHealth materials (e.g., a tailored, mobile-friendly website and text messages) to promote the correct and consistent use of size-appropriate child passenger restraints (car seats, booster seats, and seat belts). This study is designed as an adaptive randomized controlled trial, recruiting English and Spanish speaking caregivers of children 6 months to 10 years old.

DETAILED DESCRIPTION:
Motor vehicle collisions (MVCs) remain the leading cause of unintentional injury deaths among children in the United States (U.S.) and racial/ethnic minority children are disproportionately impacted as suboptimal child passenger safety behaviors are more prevalent in some communities. Existing universal approaches to promote child passenger safety have fallen short of ensuring that all child passengers are correctly using size-appropriate child passenger restraints according to guidelines published by the American Academy of Pediatrics and the National Highway Traffic Safety Administration. Precision prevention programs are urgently needed to improve child passenger safety behaviors among caregivers who have not been responsive to guidelines, laws, and public education campaigns. The proposed research will test the efficacy of Tiny Cargo, Big Deal/Abróchame Bien, Cuídame Bien (TCBD/ABCB), a bilingual emergency department (ED)-based precision prevention intervention grounded in Self-Determination Theory. TCBD/ABCB integrates personalized counseling based on principles of motivational interviewing (MI) and eHealth components including a tailored educational mobile-friendly website "site" and short message service (SMS) communications with the goal of improving child passenger safety. We hypothesize that by providing tailored child passenger safety education and personalized skills for restraint use in a manner that supports autonomous motivation the TCBD/ABCB intervention will be more efficacious than universal approaches (laws/guidelines) for realizing correct use of size-appropriate child passenger restraints.

ELIGIBILITY:
Child refers to the child of the caregiver (parent/legal guardian) who is being evaluated for recruitment and participation in the study.

Inclusion Criteria:

* Child is age 6 months to 10 years old at screening
* Child is seeking care in the Emergency Department (ED) for a non-critical injury or illness
* Child sought emergency or urgent care at a study site
* Caregiver/parent is the legal guardian of the child who is receiving or received emergency or urgent care at a study site
* Child is less than 55 inches tall
* Caregiver speaks English or Spanish
* Caregiver is 18 years old or older
* Caregiver screening survey responses indicate: child travels at least once per week in a passenger vehicle
* AND child is able to use a standard car seat or booster seat (child restraint system) but is not using an age and size-appropriate child restraint system OR travels unrestrained OR sits in the vehicle front seat OR caregiver plans to stop using the age and size-appropriate restraint in the next 6 months (planned premature transition)

Exclusion Criteria:

* Caregiver does not understand/speak English or Spanish
* Child is seeking/sought care for child abuse/neglect
* Child is seeking/sought care that requires intensive psychosocial services
* Child is seeking/sought treatment for a motor vehicle related injury
* Child is too tall for study (height = >55 inches tall)
* Caregiver is under 18 years of age
* Caregiver does not have a smart phone
* Caregiver lives outside of the state of Illinois
* Caregiver is already enrolled in this study
* Caregiver completed the screen to determine eligibility for study in the past 6 months

Exclusions applied only to in-person recruitment in the ED:

* Child is seeking treatment for a new long-term diagnosis
* Child has anticipated need for admission
* Child is seeking care for a critical illness or injury

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 513 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Macy, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results, the study protocol, statistical analysis plan, and informed consent forms will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Macy ML, Pollock B, Kendi S, Goldstick J, Cieslak K, Carter PM, Resnicow K. Multimodal Intervention and Child Passenger Safety Guideline Adherence in Young Children: A Sequential, Multiple-Assignment, Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2533912. doi: 10.1001/jamanetworkopen.2025.33912. PMID 41021229
- [Derived] Macy ML, Carter P, Kendi S, Pollock B, San Miguel L, Goldstick J, Resnicow K. "Tiny Cargo, Big Deal! Abrochame Bien, Cuidame Bien", an emergency department-based intervention to promote child passenger safety: Protocol for an adaptive randomized trial among caregivers of 6-month through 10-year-old children. Contemp Clin Trials. 2022 Sep;120:106863. doi: 10.1016/j.cct.2022.106863. Epub 2022 Jul 30. PMID 35918028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment conducted in person, 2/5/2020-3/9/2020, in a single children's hospital emergency department followed by remote recruitment, 6/29/2020-9/19/2022, in the children's hospital emergency department, two children's hospital urgent care locations, and an affiliated community hospital emergency department in metropolitan Chicago.
Pre-assignment Details: 31 caregivers were enrolled in the study and did not complete the baseline survey. Randomization occurred after completion of the baseline survey and therefore this group was not randomized. These caregivers did not participate in study activities after informed consent. 8 caregivers were determined to be ineligible after baseline survey and randomization.
Groups:
- Phases 1 and 2: Enhanced Usual Care: Participants were randomized in a 1:3 ratio (1 enhanced usual care : 3 basic intervention group) after completion of the baseline survey and received a basic information sheet (print or electronic).
  Months 1-12: Participants received eight unscheduled requests, roughly monthly, to submit photographs as their child usually travels. Feedback was provided only if critical errors and misuse were observed. Outcomes were assessed at 6 and 12 months.
- Phases 1 and 2: Basic Intervention: Tiny Cargo, Big Deal/Abróchame Bien, Cuídame Bien (TCBD/ABCB) Basic Intervention is a bilingual precision prevention intervention grounded in Self-Determination Theory. The Basic TCBD/ABCB intervention integrates one remote, personalized counseling session based on principles of motivational interviewing (MI) and mHealth components including a tailored, mobile-friendly, educational website and tailored educational and motivational short message service (SMS) text message communications sent twice each month.
  Months 1-6: Participants received four unscheduled requests to submit photographs as their child usually travels and were provided tailored feedback restraint use.
  Phase 1 Outcomes were assessed at 6 months. Participants who were guideline adherent at 6-months continued with basic mHealth. Re-randomization occurred at 6 month follow-up in a 1:1 ratio among participants who had not adopted guideline adherent behavior or still planned premature transition.
  Months 7-12: Participants who were guideline adherent at 6-months received four unscheduled requests to submit photographs as their child usually travels and were provided tailored feedback on restraint use.
  Phase 2 Outcomes were assessed at 12 months.
- Phase 2: Re-Randomized to Continue Basic Intervention (mHealth): After completion of their 6 month follow-up, participants who were re-randomized to continue the Basic (mHealth) Intervention maintained access to the tailored, mobile-friendly, educational website and tailored educational and continued to receive motivational short message service (SMS) text message communications sent twice each month. In months 7-12, this group also received four unscheduled requests to submit photographs as their child usually travels and were provided tailored feedback on restraint use. Phase 2 Outcomes were assessed at 12 months.
- Phase 2: Re-Randomized to Enhanced Intervention (Booster MI Session): After completion of 6 month follow-up, participants who were re-randomized to the Enhanced Intervention received an additional MI-based counseling session (in Months 7/8) and two additional tailored educational and motivational text messages per month (Months 7-12). Basic Intervention mHealth components for months 7-12 were continued, including photograph submission requests and feedback. Phase 2 Outcomes were assessed at 12 months.
Period: Phase 1: Baseline Intervention
Arm/Group | Phases 1 and 2: Enhanced Usual Care | Phases 1 and 2: Basic Intervention | Phase 2: Re-Randomized to Continue Basic Intervention (mHealth) | Phase 2: Re-Randomized to Enhanced Intervention (Booster MI Session)
Started | 132 | 342 | 0 | 0
Completed | 118 | 274 | 0 | 0
Not Completed | 14 | 68 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 19 | 0 | 0
Not completed — Lost to Follow-up | 11 | 49 | 0 | 0
Period: Phase 2: Rerandomized at 6 Months
Arm/Group | Phases 1 and 2: Enhanced Usual Care | Phases 1 and 2: Basic Intervention | Phase 2: Re-Randomized to Continue Basic Intervention (mHealth) | Phase 2: Re-Randomized to Enhanced Intervention (Booster MI Session)
Started | 118 | 89 | 92 | 93
Completed | 111 | 77 | 84 | 87
Not Completed | 7 | 12 | 8 | 6
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2
Not completed — Lost to Follow-up | 7 | 11 | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: Enhanced Usual Care: Participants were randomized after completion of the baseline survey and received a basic information sheet (print or electronic).
  Months 1-12: Participants received eight unscheduled requests, roughly monthly, to submit photographs as their child usually travels. Feedback was provided only if critical errors and misuse were observed. Phase 1 Outcomes were assessed at 6 months.
- Phase 1: Basic Intervention: Tiny Cargo, Big Deal/Abróchame Bien, Cuídame Bien (TCBD/ABCB) Basic Intervention is a bilingual precision prevention intervention grounded in Self-Determination Theory. The TCBD/ABCB intervention integrated one remote, personalized counseling session based on principles of motivational interviewing (MI) and mHealth components including a tailored, mobile-friendly, educational website and tailored educational and motivational short message service (SMS) text message communications sent twice each month.
  Months 1-6: Participants received four unscheduled requests to submit photographs as their child usually travels and were provided tailored feedback restraint use.
  Outcomes were assessed at 6 months. Re-randomization occurred at 6-month follow-up among participants who had not adopted guideline adherent behavior or still planned premature transition.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Enhanced Usual Care | Phase 1: Basic Intervention | Total
Number analyzed (Participants) | 132 | 342 | 474
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [32 to 40] | 36.5 [32 to 49] | 36 [32 to 40]
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 21 | 54 | 75
  30-39 years | 76 | 188 | 264
  40-58 years | 35 | 100 | 135
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 321 | 442
  Male | 11 | 21 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black, not Hispanic/Latine | 12 | 53 | 65
  Hispanic/Latine | 60 | 128 | 188
  White, not Hispanic/Latine | 41 | 136 | 177
  Other or multiple races, not Hispanic/Latine | 19 | 25 | 44
Region of Enrollment [Number; unit: participants]
  United States | 132 | 342 | 474
Preferred Language [Count of Participants; unit: Participants]
  English | 119 | 303 | 422
  Spanish | 13 | 39 | 52
Relationship to Child [Count of Participants; unit: Participants]
  Mother | 121 | 322 | 443
  Father | 10 | 20 | 30
  Grandparent | 1 | 0 | 1
Highest Education Level Achieved [Count of Participants; unit: Participants]
  High School or less | 33 | 76 | 109
  Trade School or Associates Degree | 20 | 56 | 76
  Bachelors Degree | 43 | 85 | 128
  Graduate or Professional School | 36 | 125 | 161
Children in Household [Count of Participants; unit: Participants]
  1 Child (Study Child) | 36 | 96 | 132
  2 Children | 50 | 132 | 182
  3 Children | 33 | 86 | 119
  4 Children or more | 13 | 28 | 41
Child Age Category [Count of Participants; unit: Participants]
  6 months to <3 years | 58 | 140 | 198
  3 years to <5 years | 25 | 72 | 97
  5 years through 10 years | 49 | 130 | 179
Child Sex [Count of Participants; unit: Participants]
  Male | 78 | 202 | 280
  Female | 54 | 140 | 194
Child Race and Ethnicity [Count of Participants; unit: Participants]
  Black, not Hispanic/Latine | 11 | 50 | 61
  Hispanic/Latine | 60 | 141 | 201
  White, not Hispanic/Latine | 37 | 117 | 154
  Other or multiple races, not Hispanic/Latine | 24 | 34 | 58
Baseline Child Passenger Safety Behavior [Count of Participants; unit: Participants]
  Not using recommended child passenger restraint or rides in front seat | 94 | 247 | 341
  Planning a premature transition to a less protective restraint in the next 6 months | 38 | 95 | 133

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Guideline Adherent Child Passenger Safety Behaviors at 6 Months
Description: At the 6-month follow-up assessment, conducted remotely, we reassessed the child's restraint system use and safety behaviors. For this dichotomous outcome, caregivers were considered guideline adherent if: 1) the caregiver-reported usual restraint was age and size APPROPRIATE;* and 2) the child was reported to NEVER travel UNRESTRAINED; and 3) ALWAYS seated in the vehicle BACK SEAT.
  *weight, height, and age parameters: Rear-facing appropriate if child <40 pounds; <40 inches; up to age 3 Forward-facing appropriate if child >=22 pounds, <65 pounds; >=28 inches, <49 inches, at least 3 years old Booster appropriate if child >=40 pounds, <100 pounds; High Back >=38 inches/Backless >=43 inches; <57 inches, at least 5 years old Seat Belt alone appropriate if child >=100 pounds; at least 57 inches
Time Frame: 6-Month Assessment
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Enhanced Usual Care: Participants were randomized after completion of the baseline survey and received a basic information sheet (print or electronic).
  Months 1-6: Participants received four unscheduled requests, roughly monthly, to submit photographs as their child usually travels. Feedback was provided only if critical errors and misuse were observed. Outcomes were assessed at 6 months.
- Phase 1: Basic Intervention: Tiny Cargo, Big Deal/Abróchame Bien, Cuídame Bien (TCBD/ABCB) Intervention is a bilingual precision prevention intervention grounded in Self-Determination Theory. The Basic TCBD/ABCB intervention integrates one remote, personalized counseling session based on principles of motivational interviewing (MI) and mHealth components including a tailored, mobile-friendly, educational website and tailored educational and motivational short message service (SMS) text message communications sent 2x/month.
  Months 1-6: Participants received four unscheduled requests to submit photographs as their child usually travels and received tailored feedback.
  Outcomes were assessed at 6-month follow-up.
Arm/Group | Phase 1: Enhanced Usual Care | Phase 1: Basic Intervention
Number analyzed (Participants) | 118 | 278
Participants | 38 | 131
Statistical Analysis 1: Comparison: Phase 1: Enhanced Usual Care vs Phase 1: Basic Intervention; We hypothesized the intervention group would have greater child passenger safety guideline adherence at 6 months compared with enhanced usual care group. In planning the trial, we assumed 75% of TCBD caregivers would be re-randomized. Baseline randomization was stratified by recommended CRS (rear-facing seat, forward-facing seat, booster seat) and reason for eligibility (not using the recommended CRS at baseline or planning a premature transition in the next 6 months); Test type: Superiority; p = 0.006, Regression, Logistic — The threshold for statistical significance was p = 0.05; We conducted logistic regression adjusted for randomization strata (recommended CRS and reason for eligibility); Odds Ratio (OR) = 1.876119, 95% CI 2-sided [1.193531 to 2.949084]

2. Primary Outcome: Number of Participants With Guideline Adherent Child Passenger Safety Behaviors at 12 Months
Description: At the 12-month follow-up assessment, conducted remotely, we reassessed the child's restraint system use. For this dichotomous outcome, caregivers were considered guideline adherent if: 1) the caregiver-reported usual restraint was age and size APPROPRIATE;* and 2) the child was reported to NEVER travel UNRESTRAINED; and 3) ALWAYS seated in the vehicle BACK SEAT.
  *weight, height, and age parameters: Rear-facing appropriate if child <40 pounds; <40 inches; up to age 3 Forward-facing appropriate if child >=22 pounds, <65 pounds; >=28 inches, <49 inches, at least 3 years old Booster appropriate if child >=40 pounds, <100 pounds; High Back >=38 inches/Backless >=43 inches; <57 inches, at least 5 years old Seat Belt alone appropriate if child >=100 pounds; at least 57 inches
Time Frame: 12-Month Assessment
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2: Enhanced Usual Care: EUC Months 7-12: Participants received four unscheduled requests, roughly monthly, to submit photographs as their child usually travels. Feedback was provided only if critical errors and misuse were observed. Outcomes were assessed at 12 months.
- Phase 2: Basic Intervention Guideline Adherent at 6-month Follow-up: Months 7-12: Participants received four unscheduled requests to submit photographs as their child usually travels and were provided tailored feedback on restraint use. Outcomes were assessed at 12 months.
- Phase 2: Re-Randomized to Continue Basic Intervention (mHealth): After completion of 6-month follow-up, Intervention Group participants who were re-randomized to continue the Basic Intervention received mHealth components including access to the tailored, mobile-friendly, educational website and tailored educational and motivational short message service (SMS) text message communications sent twice each month.
  In months 7-12, this group also received four unscheduled requests to submit photographs as their child usually travels and were provided tailored feedback on restraint use. Outcomes were assessed at 12 months.
- Phase 2: Re-Randomized to Enhanced Intervention (Booster MI Session): After completion of 6-month follow-up, Intervention Group participants who were re-randomized to the Enhanced Intervention received an additional MI-based counseling session (in Months 7/8) and two additional tailored educational and motivational text messages per month.
  In months 7-12, this group received Basic Intervention mHealth components, including photograph submission requests and feedback. Outcomes were assessed at 12 months.
Arm/Group | Phase 2: Enhanced Usual Care | Phase 2: Basic Intervention Guideline Adherent at 6-month Follow-up | Phase 2: Re-Randomized to Continue Basic Intervention (mHealth) | Phase 2: Re-Randomized to Enhanced Intervention (Booster MI Session)
Number analyzed (Participants) | 111 | 77 | 84 | 87
Participants | 43 | 59 | 40 | 39
Statistical Analysis 1: Comparison: Phase 2: Re-Randomized to Continue Basic Intervention (mHealth) vs Phase 2: Re-Randomized to Enhanced Intervention (Booster MI Session); This analysis is limited to the Phase 2 participants who were re-randomized at 6 months to test the hypothesis that the enhanced intervention (with booster MI session) would have greater guideline adherent child passenger safety behaviors at 12 month follow-up than the group that continued in the basic intervention (mHealth components); Test type: Superiority; p = 0.671, Regression, Logistic — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 0.8686678, 95% CI 2-sided [0.4535589 to 1.663695]
Statistical Analysis 2: Comparison: Phase 2: Enhanced Usual Care vs Phase 2: Basic Intervention Guideline Adherent at 6-month Follow-up; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.859599, 95% CI 2-sided [3.173121 to 14.82896]

3. Other Pre Specified Outcome: CPaSS Trajectories
Description: We will use latent growth curve models to identify characteristic trajectories for Child Passenger Safety Scores based on photographs of children as they typically travel obtained at baseline, months 1-4, 6-month assessment, months 8-11, and 12-month assessment.
Time Frame: 12-Month Assessment
Reporting Status: Not Posted, anticipated posting 2025-07

4. Other Pre Specified Outcome: Child Passenger Safety Score (CPaSS)
Description: At the 12-month follow-up assessment, we obtained photographs from the caregiver remotely or by research staff in-person. Photographs will be reviewed using the Child Passenger Safety Score checklist. Points will be deducted from a perfect score of 100 based on observe errors and misuse.
Time Frame: 12-Month Assessment
Reporting Status: Not Posted, anticipated posting 2025-07

5. Post Hoc Outcome: Number of Participants With Age- and Size-Appropriate Child Passenger Restraint System Use at 6 Months
Description: At the 6-month follow-up assessment, conducted remotely, we reassessed the child's restraint system use. For this dichotomous outcome, caregivers were considered guideline adherent if the caregiver-reported usual restraint was appropriate for the child's weight, height, and age.*
  *weight, height, and age parameters: Rear-facing appropriate if child <40 pounds; <40 inches; up to age 3 Forward-facing appropriate if child >=22 pounds, <65 pounds; >=28 inches, <49 inches, at least 3 years old Booster appropriate if child >=40 pounds, <100 pounds; High Back >=38 inches/Backless >=43 inches; <57 inches, at least 5 years old Seat Belt alone appropriate if child >=100 pounds; at least 57 inches
Time Frame: 6-Month Assessment
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Enhanced Usual Care: Participants were randomized in a 1:3 ratio (1 enhanced usual care : 3 basic intervention group) after completion of the baseline survey and received a basic information sheet (print or electronic).
  Months 1-6: Participants received four unscheduled requests, roughly monthly, to submit photographs as their child usually travels. Feedback was provided only if critical errors and misuse were observed. Outcomes were assessed at 6 months.
- Phase 1: Basic Intervention: Tiny Cargo, Big Deal/Abróchame Bien, Cuídame Bien (TCBD/ABCB) Basic Intervention is a bilingual precision prevention intervention grounded in Self-Determination Theory. The Basic TCBD/ABCB intervention integrates one remote, personalized counseling session based on principles of motivational interviewing (MI) and mHealth components including a tailored, mobile-friendly, educational website and tailored educational and motivational short message service (SMS) text message communications sent twice each month.
  Months 1-6: Participants received four unscheduled requests to submit photographs as their child usually travels and were provided tailored feedback restraint use. Outcomes were assessed at 6 months.
Arm/Group | Phase 1: Enhanced Usual Care | Phase 1: Basic Intervention
Number analyzed (Participants) | 118 | 278
Participants | 52 | 156
Statistical Analysis 1: Comparison: Phase 1: Enhanced Usual Care vs Phase 1: Basic Intervention; Test type: Superiority; p = 0.032, Regression, Logistic — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 1.74029, 95% CI 2-sided [1.049169 to 2.886676]

6. Post Hoc Outcome: Number of Participants With Age- and Size-Appropriate Child Passenger Restraint System Use at 12 Months
Description: At the 12-month follow-up assessment, conducted remotely, we reassessed the child's restraint system use and safety behaviors. For this dichotomous outcome, caregivers were considered guideline adherent if the caregiver-reported usual restraint was appropriate for the child's weight, height, and age.*
  *weight, height, and age parameters: Rear-facing appropriate if child <40 pounds; <40 inches; up to age 3 Forward-facing appropriate if child >=22 pounds, <65 pounds; >=28 inches, <49 inches, at least 3 years old Booster appropriate if child >=40 pounds, <100 pounds; High Back >=38 inches/Backless >=43 inches; <57 inches, at least 5 years old Seat Belt alone appropriate if child >=100 pounds; at least 57 inches
Time Frame: 12-Month Assessment
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2: Basic Intervention Guideline Adherent at 6-month Follow-up: Caregivers with guideline adherence at 6 month follow-up were not re-randomized.
  Months 7-12: Participants maintained access to the mHealth components of the basic intervention and received four unscheduled requests to submit photographs as their child usually travels and were provided tailored feedback on restraint use. Outcomes were assessed at 12 months.
- Phase 2: Re-Randomized to Basic Intervention: After completion of 6-month follow-up, Intervention Group participants who were re-randomized to continue the Basic Intervention received mHealth components including access to the tailored, mobile-friendly, educational website and tailored educational and motivational short message service (SMS) text message communications sent twice each month.
  In months 7-12, this group also received four unscheduled requests to submit photographs as their child usually travels and were provided tailored feedback on restraint use. Outcomes were assessed at 12 months.
- Phase 2: Re-Randomized to Enhanced Intervention: After completion of 6-month follow-up, Intervention Group participants who were re-randomized to the Enhanced Intervention received an additional MI-based counseling session (in Months 7/8) and two additional tailored educational and motivational text messages per month.
  In months 7-12, this group received Basic Intervention mHealth components, including photograph submission requests and feedback. Outcomes were assessed at 12 months.
Arm/Group | Phase 2: Enhanced Usual Care | Phase 2: Basic Intervention Guideline Adherent at 6-month Follow-up | Phase 2: Re-Randomized to Basic Intervention | Phase 2: Re-Randomized to Enhanced Intervention
Number analyzed (Participants) | 111 | 77 | 84 | 87
Participants | 59 | 65 | 46 | 49
Statistical Analysis 1: Comparison: Phase 2: Re-Randomized to Basic Intervention vs Phase 2: Re-Randomized to Enhanced Intervention; Test type: Superiority; p = 0.752, Regression, Logistic — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 1.112874, 95% CI 2-sided [0.5735782 to 2.159233]
Statistical Analysis 2: Comparison: Phase 2: Enhanced Usual Care vs Phase 2: Basic Intervention Guideline Adherent at 6-month Follow-up; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.959981, 95% CI 2-sided [3.321933 to 19.07362]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year.
Groups:
- Phase 1: Enhanced Usual Care (EUC): Participants randomized to EUC received a basic information sheet (print or electronic) at enrollment.
  EUC Months 1-6: Participants received four unscheduled requests, roughly monthly, to submit photographs as their child usually travels. Feedback was provided only if critical errors and misuse were observed. Outcomes were assessed at 6 months.
- Phase 1: Intervention: Tiny Cargo, Big Deal/Abróchame Bien, Cuídame Bien (TCBD/ABCB) Basic Intervention is a bilingual precision prevention intervention grounded in Self-Determination Theory. The TCBD/ABCB intervention integrated one remote, personalized counseling session based on principles of motivational interviewing (MI) and mHealth components including a tailored, mobile-friendly, educational website and tailored educational and motivational short message service (SMS) text message communications sent twice each month.
  Months 1-6: Participants received four unscheduled requests to submit photographs as their child usually travels and were provided tailored feedback restraint use.
  Outcomes were assessed at 6 months. Re-randomization occurred at 6-month follow-up among participants who had not adopted guideline adherent behavior or still planned premature transition.
- Phase 2: Enhanced Usual Care (EUC): EUC Months 7-12: Participants received four unscheduled requests, roughly monthly, to submit photographs as their child usually travels. Feedback was provided only if critical errors and misuse were observed. Outcomes were assessed at 12 months.
- Phase 2: Guideline Adherent at 6-month Follow-up: Months 7-12: Participants received four unscheduled requests to submit photographs as their child usually travels and were provided tailored feedback on restraint use. Outcomes were assessed at 12 months.
Arm/Group | Phase 1: Enhanced Usual Care (EUC) | Phase 1: Intervention | Phase 2: Enhanced Usual Care (EUC) | Phase 2: Guideline Adherent at 6-month Follow-up | Phase 2: Re-Randomized to Continue Basic Intervention (mHealth) | Phase 2: Re-Randomized to Enhanced Intervention (Booster MI Session)
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/274 | 0/111 | 0/77 | 0/84 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/274 | 0/111 | 0/77 | 0/84 | 0/87
Other Adverse Events (participants affected / at risk) | 2/118 | 7/274 | 1/111 | 3/77 | 2/84 | 4/87
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Enhanced Usual Care (EUC) (N=118) | Phase 1: Intervention (N=274) | Phase 2: Enhanced Usual Care (EUC) (N=111) | Phase 2: Guideline Adherent at 6-month Follow-up (N=77) | Phase 2: Re-Randomized to Continue Basic Intervention (mHealth) (N=84) | Phase 2: Re-Randomized to Enhanced Intervention (Booster MI Session) (N=87)
Possible Delayed Transition (General disorders) | 2 (2) | 7 (7) | 1 (1) | 3 (3) | 2 (2) | 4 (4) — Caregiver reported child's weight or height was above the maximum weight or height for a typical child passenger restraint system (CRS) within that mode (e.g., rear-facing), which could indicate the child was too heavy or tall for their usual CRS.

LIMITATIONS AND CAVEATS:
Recruitment was negatively impacted by the coronavirus disease 19 (COVID-19) pandemic and we were unable to achieve our target sample size. The Child Passenger Safety Score (CPaSS) Tool requires additional calibration to assure greater reliability before we are able to report outcomes that are dependent upon this score.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT04238247/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT04238247/ICF_001.pdf